CLINICAL TRIAL: NCT00433914
Title: A Phase 2, Single Blind, Single Center, Randomized Study of the Safety, Tolerability and Immunogenicity of Novartis Meningococcal B Recombinant Vaccine +/- OMV, When Administered to Healthy Infants 6-8 Months Old
Brief Title: Safety, Tolerability and Immunogenicity of Two Different Formulations of Meningococcal B Recombinant Vaccine, When Administered to Healthy Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V72P9; Eudract Number: 2006-005589-38
Record Dates: First submitted 2007-02-09; First posted 2007-02-12 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Meningococcal Disease
Keywords: Meningococcal disease, prevention, vaccination
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- rMenB (Experimental): 6-8 months-old infants received 3 doses of rMenB vaccine without OMV-NZ at 6-8 months of age, 2 months later and 12 months of age.
  Interventions: Biological: rMenB
- rMenB+OMV (Experimental): 6-8 months-old infants received 3 doses of rMenB vaccine with OMV-NZ at 6-8 months of age, 2 months later and 12 months of age.
  Interventions: Biological: rMenB+OMV

INTERVENTIONS:
Biological: rMenB — One dose (0.5 mL) of rMenB vaccine without OMV-NZ supplied as a full liquid formulation in a prefilled syringe was administered into the anterolateral area of the right thigh.
  Other Names: Serogroup B meningococcal recombinant vaccine without OMV-NZ
  Arms: rMenB
Biological: rMenB+OMV — One dose (0.5 mL) of rMenB vaccine with OMV-NZ supplied as a full liquid formulation in a prefilled syringe was administered into the anterolateral area of the right thigh.
  Other Names: Serogroup B meningococcal recombinant vaccine with OMV-NZ
  Arms: rMenB+OMV

SUMMARY:
To explore safety, Tolerability and immunogenicity of two formulations of a Meningococcal B Recombinant Vaccine when administered to healthy infants.

ELIGIBILITY:
Inclusion Criteria:

* healthy 6-8 months old infants

Exclusion Criteria:

* previous receipt of any meningococcal B vaccine;
* previous ascertained or suspected disease caused by N meningitidis;
* history of any anaphylactic shock, asthma, urticaria or other allergic reaction after previous vaccinations or known hypersensitivity to any vaccine component;
* any present or suspected serious acute or chronic disease
* known or suspected autoimmune disease or impairment /alteration of immune function

Ages: 6 Months to 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2007-02; Primary Completion 2007-12 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines (formerly Chiron Vaccines) Novartis, Study Chair — Novartis Vaccines
Locations (1):
- Oxford, United Kingdom

REFERENCES:
- [Derived] Viviani V, Biolchi A, Pizza M. Synergistic activity of antibodies in the multicomponent 4CMenB vaccine. Expert Rev Vaccines. 2022 May;21(5):645-658. doi: 10.1080/14760584.2022.2050697. Epub 2022 Mar 14. PMID 35257644
- [Derived] Snape MD, Dawson T, Oster P, Evans A, John TM, Ohene-Kena B, Findlow J, Yu LM, Borrow R, Ypma E, Toneatto D, Pollard AJ. Immunogenicity of two investigational serogroup B meningococcal vaccines in the first year of life: a randomized comparative trial. Pediatr Infect Dis J. 2010 Nov;29(11):e71-9. doi: 10.1097/INF.0b013e3181f59f6d. PMID 20844462

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at one study center in the United Kingdom (UK).
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- rMenB: 6-8 month-old infants received 3 doses of rMenB vaccine without OMV-NZ at 6-8 months of age, 2 months later and at 12 months of age.
- rMenB+OMV: 6-8 month-old infants received 3 doses of rMenB vaccine with OMV-NZ at 6-8 months of age, 2 months later and at 12 months of age.
Period: Overall Study
Arm/Group | rMenB | rMenB+OMV
Started | 30 | 30
Completed | 30 | 27
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | rMenB | rMenB+OMV | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: Months] | 7.0 (0.8) | 7.1 (0.7) | 7.1 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 18 | 32
  Male | 16 | 12 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Bactericidal Titers ≥1:4 Against Meningococcal Strains One Month After Second and Third Vaccination of rMenB Vaccine With and Without OMV-NZ
Description: Immunogenicity was measured as the percentage of subjects who achieved bactericidal titers ≥1:4 against meningococcal strains 44/76-SL, 5/99, NZ98/254 (major strains), UK P1.7-2,4, GB101, GB355 and GB364 (additional strains), evaluated using serum bactericidal assay, before vaccination (baseline) and one month after second vaccination (2 months later after vaccination at 6-8 months of age) and third vaccination (at 12 months of age).
Time Frame: Baseline and one month after second and third vaccination
Population: Analysis was performed on the per protocol (PP) population set, i.e. all subjects in the enrolled population who received all the relevant doses of vaccine correctly; provided evaluable serum samples at the relevant time points; and had no major protocol violation as defined prior to analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB | rMenB+OMV
Number analyzed (Participants) | 25 | 24
Percentage of subjects
  Strain 44/76-SL - Baseline | 8 [1 to 26] | 29 [13 to 51]
  Strain 44/76-SL - Post-2nd Vaccination (N=25,23) | 100 [86 to 100] | 100 [85 to 100]
  Strain 44/76-SL - Post-3rd Vaccination (N=24,24) | 100 [86 to 100] | 100 [86 to 100]
  Strain 5/99 - Baseline | 0 [0 to 14] | 0 [0 to 14]
  Strain 5/99 - Post-2nd Vaccination (N=25,23) | 100 [86 to 100] | 100 [85 to 100]
  Strain 5/99 - Post-3rd Vaccination (N=24,24) | 100 [86 to 100] | 100 [86 to 100]
  Strain NZ98/254 - Baseline | 0 [0 to 14] | 0 [0 to 14]
  Strain NZ98/254 - Post-2nd Vaccination (N=24,22) | 4 [0 to 21] | 95 [77 to 100]
  Strain NZ98/254 - Post-3rd Vaccination (N=22,24) | 9 [1 to 29] | 96 [79 to 100]
  Strain UK P1.7-2,4 - Baseline (N=24,21) | 0 [0 to 14] | 0 [0 to 16]
  Strain UKP1.7-2,4 - Post-2nd Vaccination (N=23,19) | 0 [0 to 15] | 100 [82 to 100]
  Strain UKP1.7-2,4 - Post-3rd Vaccination (N=21,22) | 5 [0 to 24] | 100 [85 to 100]
  Strain GB101 - Baseline (N=24,21) | 0 [0 to 14] | 10 [1 to 30]
  Strain GB101 - Post-2nd Vaccination (N=22,21) | 23 [8 to 45] | 67 [43 to 85]
  Strain GB101 - Post-3rd Vaccination (N=22,22) | 27 [11 to 50] | 73 [50 to 89]
  Strain GB355 - Baseline (N=12,11) | 0 [0 to 26] | 0 [0 to 28]
  Strain GB355 - Post-2nd Vaccination (N=11,14) | 0 [0 to 28] | 7 [0 to 34]
  Strain GB355 - Post-3rd Vaccination (N=12,11) | 0 [0 to 26] | 18 [2 to 52]
  Strain GB364 - Baseline (N=22,17) | 9 [1 to 29] | 12 [1 to 36]
  Strain GB364 - Post-2nd Vaccination (N=19,16) | 95 [74 to 100] | 88 [62 to 98]
  Strain GB364 - Post-3rd Vaccination (N=17,19) | 88 [64 to 99] | 95 [74 to 100]

2. Primary Outcome: Percentage of Subjects With Bactericidal Titers ≥1:8 Against Meningococcal Strains One Month After Second and Third Vaccination of rMenB Vaccine With and Without OMV-NZ
Description: Immunogenicity was measured as the percentage of subjects who achieved bactericidal titers ≥1:8 against meningococcal strains 44/76-SL, 5/99, NZ98/254 (major strains), UK P1.7-2,4, GB101, GB355 and GB364 (additional strains), before vaccination (baseline) and one month after second vaccination (2 months after vaccination at 6-8 months) and third vaccination (at 12 months of age).
Time Frame: Baseline and one month after second and third vaccination
Population: Analysis was performed on the per protocol (PP) population set.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB | rMenB+OMV
Number analyzed (Participants) | 25 | 24
Percentage of subjects
  Strain 44/76-SL - Baseline | 0 [0 to 14] | 4 [0 to 21]
  Strain 44/76-SL - Post-2nd Vaccination (N=25,23) | 96 [80 to 100] | 100 [85 to 100]
  Strain 44/76-SL - Post-3rd Vaccination (N=24,24) | 100 [86 to 100] | 100 [86 to 100]
  Strain 5/99 - Baseline | 0 [0 to 14] | 0 [0 to 14]
  Strain 5/99 - Post-2nd Vaccination (N=25,23) | 100 [86 to 100] | 100 [85 to 100]
  Strain 5/99 - Post-3rd Vaccination (N=24,24) | 100 [86 to 100] | 100 [86 to 100]
  Strain NZ98/254 - Baseline | 0 [0 to 14] | 0 [0 to 14]
  Strain NZ98/254 - Post-2nd Vaccination (N=24,22) | 0 [0 to 14] | 91 [71 to 99]
  Strain NZ98/254 - Post-3rd Vaccination (N=22,24) | 5 [0 to 23] | 96 [79 to 100]
  Strain UK P1.7-2,4 - Baseline (N=24,21) | 0 [0 to 14] | 0 [0 to 16]
  Strain UKP1.7-2,4 - Post-2nd Vaccination (N=23,19) | 0 [0 to 15] | 84 [60 to 97]
  Strain UKP1.7-2,4 - Post-3rd Vaccination (N=21,22) | 0 [0 to 16] | 95 [77 to 100]
  Strain GB101 - Baseline (N=24,21) | 0 [0 to 14] | 10 [1 to 30]
  Strain GB101 - Post-2nd Vaccination (N=22,21) | 9 [1 to 29] | 33 [15 to 57]
  Strain GB101 - Post-3rd Vaccination (N=22,22) | 14 [3 to 35] | 45 [24 to 68]
  Strain GB355 - Baseline (N=12,11) | 0 [0 to 26] | 0 [0 to 28]
  Strain GB355 - Post-2nd Vaccination (N=11,14) | 0 [0 to 28] | 0 [0 to 23]
  Strain GB355 - Post-3rd Vaccination (N=12,11) | 0 [0 to 26] | 0 [0 to 28]
  Strain GB364 - Baseline (N=22,17) | 0 [0 to 15] | 0 [0 to 20]
  Strain GB364 - Post-2nd Vaccination (N=19,16) | 74 [49 to 91] | 69 [41 to 89]
  Strain GB364 - Post-3rd Vaccination (N=17,19) | 71 [44 to 90] | 84 [60 to 97]

3. Secondary Outcome: Percentage of Subjects With Four-fold Rise in Bactericidal Titers Against Meningococcal Strains One Month After Second and Third Vaccination of rMenB Vaccine With and Without OMV-NZ
Description: Immunogenicity was measured as the percentage of subjects who achieved a four-fold increase in bactericidal titers against meningococcal strains 44/76-SL, 5/99, NZ98/254 (major strains), UK P1.7-2,4, GB101, GB355 and GB364 (additional strains), one month after second vaccination (2 months after vaccination at 6-8 months) and third vaccination (at 12 months of age).
Time Frame: One month after second and third vaccination
Population: Analysis was performed on the per protocol (PP) population set.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB | rMenB+OMV
Number analyzed (Participants) | 25 | 24
Percentage of subjects
  Strain 44/76-SL - Post-2nd Vaccination (N=25,23) | 96 [80 to 100] | 100 [85 to 100]
  Strain 44/76-SL - Post-3rd Vaccination (N=24,24) | 100 [86 to 100] | 100 [86 to 100]
  Strain 5/99 - Post-2nd Vaccination (N=25,23) | 100 [86 to 100] | 100 [85 to 100]
  Strain 5/99 - Post-3rd Vaccination | 100 [86 to 100] | 100 [86 to 100]
  Strain NZ98/254 - Post-2nd Vaccination (N=24,22) | 0 [0 to 14] | 91 [71 to 99]
  Strain NZ98/254 - Post-3rd Vaccination (N=22,24) | 5 [0 to 23] | 96 [79 to 100]
  Strain UKP1.7-2,4 - Post-2nd Vaccination (N=22,17) | 0 [0 to 15] | 88 [64 to 99]
  Strain UKP1.7-2,4 - Post-3rd Vaccination (N=20,20) | 0 [0 to 17] | 95 [75 to 100]
  Strain GB101 - Post-2nd Vaccination (N=21,18) | 10 [1 to 30] | 22 [6 to 48]
  Strain GB101 - Post-3rd Vaccination (N=21,19) | 14 [3 to 36] | 32 [13 to 57]
  Strain GB355 - Post-2nd Vaccination (N=5,7) | 0 [0 to 52] | 0 [0 to 41]
  Strain GB355 - Post-3rd Vaccination (N=7,6) | 0 [0 to 41] | 0 [0 to 46]
  Strain GB364 - Post-2nd Vaccination (N=17,14) | 76 [50 to 93] | 64 [35 to 87]
  Strain GB364 - Post-3rd Vaccination (N=15,15) | 80 [52 to 96] | 80 [52 to 96]
  287-953proteinantigen-Post-2ndVaccination(N=25,23) | 100 [86 to 100] | 100 [85 to 100]
  287-953proteinantigen-Post-3rdVaccination(N=24,25) | 100 [86 to 100] | 100 [86 to 100]

4. Secondary Outcome: Geometric Mean Bactericidal Titers Against Meningococcal Strains One Month After Second and Third Vaccination of rMenB Vaccine With and Without OMV-NZ
Description: The immune response was measured as the geometric mean bactericidal titers directed against meningococcal strains 44/76-SL, 5/99, NZ98/254 (major strains), UK P1.7-2,4, GB101, GB355 and GB364 (additional strains), before vaccination (baseline) and one month after second vaccination (2 months after vaccination at 6-8 months) and third vaccination (at 12 months of age).
Time Frame: Baseline and one month after second and third vaccination
Population: Analysis was performed on the per protocol (PP) population set.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean titers
Arm/Group | rMenB | rMenB+OMV
Number analyzed (Participants) | 25 | 24
Geometric mean titers
  Strain 44/76-SL - Baseline | 1.16 [0.89 to 1.52] | 1.70 [1.29 to 2.24]
  Strain 44/76-SL - Post-2nd Vaccination (N=25,23) | 94 [66 to 134] | 250 [173 to 361]
  Strain 44/76-SL - Post-3rd Vaccination (N=24,24) | 109 [79 to 153] | 189 [136 to 263]
  Strain 5/99 - Baseline | 1.00 [0.94 to 1.07] | 1.05 [0.98 to 1.12]
  Strain 5/99 - Post-2nd Vaccination (N=25,23) | 710 [532 to 947] | 534 [395 to 721]
  Strain 5/99 - Post-3rd Vaccination (N=24,24) | 1202 [929 to 1555] | 906 [700 to 1172]
  Strain NZ98/254 - Baseline | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Strain NZ98/254 - Post-2nd Vaccination (N=24,22) | 1.06 [0.82 to 1.38] | 27 [21 to 36]
  Strain NZ98/254 - Post-3rd Vaccination (N=22,24) | 1.21 [0.86 to 1.72] | 44 [32 to 62]
  Strain UK P1.7-2,4 - Baseline (N=24,21) | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Strain UKP1.7-2,4 - Post-2nd Vaccination (N=23,19) | 1.00 [0.75 to 1.34] | 17 [12 to 24]
  Strain UKP1.7-2,4 - Post-3rd Vaccination (N=21,22) | 1.07 [0.72 to 1.58] | 34 [23 to 50]
  Strain GB101 - Baseline (N=24,21) | 1.12 [0.81 to 1.56] | 1.49 [1.05 to 2.11]
  Strain GB101 - Post-2nd Vaccination (N=22,21) | 1.82 [1.14 to 2.90] | 4.56 [2.83 to 7.35]
  Strain GB101 - Post-3rd Vaccination (N=22,22) | 2.20 [1.14 to 4.23] | 9.36 [4.87 to 18]
  Strain GB355 - Baseline (N=12,11) | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Strain GB355 - Post-2nd Vaccination (N=11,14) | 1.00 [0.83 to 1.21] | 1.16 [0.98 to 1.37]
  Strain GB355 - Post-3rd Vaccination (N=12,11) | 1.06 [0.82 to 1.36] | 1.46 [1.12 to 1.90]
  Strain GB364 - Baseline (N=22,17) | 1.46 [1.19 to 1.79] | 1.50 [1.19 to 1.90]
  Strain GB364 - Post-2nd Vaccination (N=19,16) | 11 [6.39 to 19] | 12 [6.75 to 23]
  Strain GB364 - Post-3rd Vaccination (N=17,19) | 12 [6.17 to 22] | 21 [11 to 37]

5. Secondary Outcome: Geometric Mean ELISA Concentration Against Meningococcal 287-953 Antigen One Month After Second and Third Vaccination of rMenB Vaccine With and Without OMV-NZ
Description: The immune response was measured as the geometric mean concentrations (GMCs) against the meningococcal antigen 287-953, evaluated using enzyme-linked immunosorbent assay (ELISA), before vaccination (baseline) and one month after second vaccination (2 months after vaccination at 6-8 months) and third vaccination (at 12 months of age).
Time Frame: Baseline and one month after second and third vaccination
Population: Analysis was performed on the per protocol (PP) population set.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | rMenB | rMenB+OMV
Number analyzed (Participants) | 25 | 25
µg/mL
  Antigen 287-953 - Baseline | 24 [21 to 28] | 21 [18 to 24]
  Antigen 287-953 - Post-2nd Vaccination (N=25,23) | 1759 [1331 to 2324] | 2912 [2178 to 3894]
  Antigen 287-953 - Post-3rd Vaccination (N=24,25) | 2298 [1778 to 2970] | 3521 [2739 to 4527]

6. Secondary Outcome: Percentage of Subjects With Four-fold Rise in ELISA Concentration Against Meningococcal 287-953 Antigen One Month After Second and Third Vaccination of rMenB Vaccine With and Without OMV-NZ
Description: Immunogenicity was measured as the percentage of subjects who achieved a four-fold increase in ELISA geometric mean concentrations against meningococcal 287-953 antigen, one month after second vaccination (2 months after vaccination at 6-8 months) and third vaccination (at 12 months of age).
Time Frame: One month after second and third vaccination
Population: Analysis was performed on the per protocol (PP) population set.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB | rMenB+OMV
Number analyzed (Participants) | 25 | 25
Percentage of subjects
  Antigen 287-953 - Post-2nd Vaccination (N=25,23) | 100 [86 to 100] | 100 [85 to 100]
  Antigen 287-953 - Post-3rd Vaccination (N=24,25) | 100 [86 to 100] | 100 [86 to 100]

7. Secondary Outcome: Number of Subjects Who Reported Solicited Local and Systemic Reactions After Each Vaccination of rMenB Vaccine With and Without OMV-NZ
Description: Safety was assessed as the number of subjects who reported solicited local and systemic reactions from day 1 through day 7 after each vaccination of rMenB vaccine with and without OMV-NZ administered at 6-8 months (vaccination 1), 2 months later (vaccination 2) and at 12 months (vaccination 3).
Time Frame: Day 1 through day 7 after each vaccination
Population: Analysis was performed on the safety set, i.e. all subjects in the exposed population who provided post-baseline safety data.
Measure: Number; unit: Number of subjects
Arm/Group | rMenB | rMenB+OMV
Number analyzed (Participants) | 30 | 30
Number of subjects
  Local reactions | 29 | 29
  Tenderness - Vaccination 1 | 4 | 9
  Tenderness - Vaccination 2 (N=30,28) | 5 | 11
  Tenderness - Vaccination 3 (N=30,27) | 12 | 10
  Erythema - Vaccination 1 | 26 | 26
  Erythema - Vaccination 2 (N=30,28) | 22 | 25
  Erythema - Vaccination 3 (N=30,27) | 24 | 26
  Induration - Vaccination 1 | 15 | 18
  Induration - Vaccination 2 (N=30,28) | 12 | 16
  Induration - Vaccination 3 (N=30,27) | 15 | 18
  Swelling - Vaccination 1 | 4 | 11
  Swelling - Vaccination 2 (N=30,28) | 9 | 10
  Swelling - Vaccination 3 (N=30,27) | 11 | 9
  Systemic reactions | 22 | 28
  Change in eating habits - Vaccination 1 (N=30,29) | 6 | 8
  Change in eating habits - Vaccination 2 (N=30,27) | 1 | 7
  Change in eating habits - Vaccination 3 (N=30,27) | 8 | 5
  Sleepiness - Vaccination 1 | 7 | 11
  Sleepiness - Vaccination 2 (N=30,28) | 7 | 8
  Sleepiness - Vaccination 3 (N=30,27) | 7 | 4
  Vomiting - Vaccination 1 | 6 | 4
  Vomiting - Vaccination 2 (N=30,28) | 1 | 3
  Vomiting - Vaccination 3 (N=30,27) | 6 | 2
  Diarrhea - Vaccination 1 | 2 | 5
  Diarrhea - Vaccination 2 (N=30,28) | 4 | 1
  Diarrhea - Vaccination 3 (N=30,27) | 5 | 5
  Unusual crying - Vaccination 1 | 2 | 3
  Unusual crying - Vaccination 2 (N=30,28) | 2 | 2
  Unusual crying - Vaccination 3 (N=30,27) | 4 | 7
  Irritability - Vaccination 1 | 14 | 14
  Irritability - Vaccination 2 (N=30,28) | 10 | 17
  Irritability - Vaccination 3 (N=30,28) | 13 | 18
  Rash - Vaccination 1 | 3 | 3
  Rash - Vaccination 2 (N=30,28) | 5 | 4
  Rash - Vaccination 3 (N=30,27) | 5 | 4
  Fever (≥38 °C) - Vaccination 1 | 1 | 3
  Fever (≥38 °C) - Vaccination 2 (N=30,28) | 2 | 3
  Fever (≥38 °C) - Vaccination 3 (N=30,27) | 4 | 1
  Analg/Antipyr medications used - Vaccination 1 | 10 | 18
  Analg/Antipyr medications used - Vaccination 2 | 12 | 17
  Analg/Antipyr medications used - Vaccination 3 | 15 | 16

ADVERSE EVENTS:
Time Frame: Throughout the study period (day 1 to follow-up of 180 days after 12 months vaccination)
Arm/Group | rMenB | rMenB+OMV
Serious Adverse Events (participants affected / at risk) | 5/30 | 1/30
Other Adverse Events (participants affected / at risk) | 30/30 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rMenB (N=30) | rMenB+OMV (N=30)
Cellulitis (Infections and infestations) | 1 | 0
Croup infectious (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Febrile convulsion (Nervous system disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | rMenB (N=30) | rMenB+OMV (N=30)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Somnolence (Nervous system disorders) | 14 | 16
Induration (General disorders) | 1 | 4
Injection site erythema (General disorders) | 28 | 28
Injection site swelling (General disorders) | 14 | 17
Pyrexia (General disorders) | 7 | 6
Swelling (General disorders) | 0 | 3
Crying (General disorders) | 5 | 10
Injection site pain (General disorders) | 13 | 18
vaccination site erythema (General disorders) | 2 | 0
Irritability (Psychiatric disorders) | 18 | 25
Eating disorder (Psychiatric disorders) | 13 | 14
Diarrhoea (Gastrointestinal disorders) | 16 | 13
Teething (Gastrointestinal disorders) | 11 | 13
Vomiting (Gastrointestinal disorders) | 16 | 10
Eczema (Skin and subcutaneous tissue disorders) | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 8 | 9
Conjunctivitis (Infections and infestations) | 1 | 5
Gastroenteritis (Infections and infestations) | 0 | 4
Lower respiratory tract infection (Infections and infestations) | 2 | 3
Nasopharyngitis (Infections and infestations) | 1 | 3
Otitis media (Infections and infestations) | 2 | 1
Rhinitis (Infections and infestations) | 5 | 3
Tonsilitis (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Varicella (Infections and infestations) | 2 | 0
Viral rash (Infections and infestations) | 2 | 2
Viral upper respiratory tract infection (Infections and infestations) | 4 | 0
Injection site induration (General disorders) | 20 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No